CLINICAL TRIAL: NCT03544255
Title: Drug Screening of Pancreatic Cancer Organoids Developed From EUS-FNA Guided Biopsy Tissues
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ying Lv (Other)
Responsible Party: Sponsor-Investigator, Ying Lv, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Other Study IDs: EFOP-01
Record Dates: First submitted 2018-04-17; First posted 2018-06-01 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Cancer; Pancreas Adenocarcinoma
Keywords: pancreatic cancer; EUS-FNA; organoid
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will create organoids from pancreatic cancer biopsies achieved from EUS-FNA. And the pancreatic cancer organoids will be passed and frozen in standard conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Biopsy — Two extra EUS-FNA guided pancreatic biopsies collected for only research purposes.

SUMMARY:
We are going to establish "organoid" models from pancreatic cancer biopsies achieved via EUS-FNA. Then the sensitivity of the selected FDA-approved anti-cancer drugs will be tested in these organoids.

DETAILED DESCRIPTION:
The survival rate of pancreatic cancer, a kind of malignant tumor, remains poor due to lack of effective treatments. Recently, a new model called "organoid" has been generated from human and murine pancreatic cancer tissues. These organoids are developed from large pieces of surgical tissues or small biopsies taken from EUS-FNA guided samples. Here in our study we are going to establish "organoid" models from pancreatic cancer biopsies achieved via EUS-FNA. After successful generation of these organoids, we will treat them with the selected FDA-approved anti-cancer drugs, and assess the responses to these anti-cancer agents in our established organoids.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients suspected to have pancreatic cancer who will receive EUS-FNA for diagnosis; 2) Patients who have signed the informed consent.

Exclusion Criteria:

* 1) Those who are under the age of 18; 2) Patients who have received adjuvant chemoradiotherapies or other anti-tumor therapies; 3) Patients with critical illness and cannot tolerate the operations; 4) Women who have been pregnant or are planning to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected to have pancreatic cancer who are going to receive EUS-FNA operations for diagnostic purposes.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of organoids successfully generated from pancreatic cancer biopsies | 09/01/2018-06/01/2019
  Successful isolation of pancreatic cancer organoids within 2 weeks of EUS-FNA operation will be defined as successful establishment of an organoid. We will calculate the total number of organoids generated in our center.

SECONDARY OUTCOMES:
Response of the pancreatic cancer organoids to the selected anti-cancer drugs | 06/01/2019-06/01/2020
  We will treat the established organoids with the selected FDA-approved drugs. Then the anti-cancer activity of these drugs will be tested using CellTiter-Glo 3D Cell Viability Assay (Promega).

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lv, PhD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided